CLINICAL TRIAL: NCT05689931
Title: Blood Leukocyte Profiling in Eosinophilic Type 2 Asthma: Influence of Systemic IL-5 Targeting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 1072615
Record Dates: First submitted 2022-12-15; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Asthma patients initiating Mepolizumab treatment: Patients will be selected on the standard criteria used to select eligible asthma patients for mepolizumab treatment (i.e. patients with eosinophilic asthma that are not controlled by conventional high dose ICS and LABA etc). All eligible asthma patients may be included. Exclusion criteria: any infection
  Interventions: Biological: Mepolizumab; Drug: Standard inhaled corticosteroids (ICS) and long-acting beta 2 agonists (LABA)
- Asthma patients already on Mepolizumab treatment: Patients that have been selected and given Mepolizumab treatment for > 4 months according to standard eligible and treatment regimen criteria (i.e. patients with eosinophilic asthma that are not controlled by conventional high dose ICS and LABA etc). All eligible asthma patients that have been on Mepolizumab treatment for > 4 weeks will be included. Exclusion criteria: any infections
  Interventions: Biological: Mepolizumab; Drug: Standard inhaled corticosteroids (ICS) and long-acting beta 2 agonists (LABA)
- Asthma patients without Mepolizumab treatment: Inclusion: Asthma patients without any biological (antibody-based) treatment but on routine ICS and LABA treatment as part of their normal care. Exclusion criteria are any infections
  Interventions: Drug: Standard inhaled corticosteroids (ICS) and long-acting beta 2 agonists (LABA)
- Healthy non-asthmatic control subjects: Exclusion criteria: previous history of lung disease, chronic inflammatory condition, or atopy, or cardiovascular disease. Diagnosed or perceived infection within 3 weeks prior to blood sampling

INTERVENTIONS:
Biological: Mepolizumab — Mepolizumab is administered by subcutaneous injection with guideline recommended patient selection and dosing for treatment of eosinophilic asthma.
  Accordingly, the Mepolizumab treatment is given as add-on therapy to standard inhaled corticosteroids (ICS) and long-acting beta 2 agonists (LABA)
  Other Names: Mepolizumab (brand name: Nucala)
  Groups: Asthma patients already on Mepolizumab treatment; Asthma patients initiating Mepolizumab treatment
Drug: Standard inhaled corticosteroids (ICS) and long-acting beta 2 agonists (LABA) — Routine asthma treatment with inhaled corticosteroids (ICS) and long-acting beta 2 agonists (LABA)
  Other Names: ICS and LABA
  Groups: Asthma patients already on Mepolizumab treatment; Asthma patients initiating Mepolizumab treatment; Asthma patients without Mepolizumab treatment

SUMMARY:
The goal of this exploratory and observational prospective study is to study the composition and phenotypes of blood leukocytes collected from asthmatic patients before and after instantiated treatment with the interleukin-5 neutralizing antibody mepolizumab. Comparisons will be made to leukocyte profiles in patients already on mepolizumab treatment, asthma patients without any biological treatment, and non-diseased control subjects.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory and obstructive condition affecting the airways. The disease is commonly associated with elevated blood eosinophils and tissue eosinophilia. Many aspects of the pathophysiological mechanisms and clinical symptoms are controlled by conventional therapies such as inhaled corticosteroids (ICS) and long acting β2 agonists. However, some patients remain clinically uncontrolled and need additional treatment such as direct targeting of eosinophil granulocytes by neutralizing the eosinophil-promoting cytokine interleukin 5 (IL5). Mepolizumab is a humanized monoclonal IL-5 neutralizing antibody that is used to treat patients with moderate-severe eosinophilic asthma. While a marked reduction of eosinophils is a key effect of mepolizumab, the exact mechanism of action is unknown. Apart from basophils, that also express the receptor for IL-5, other leukocytes are likely to be indirectly affected by the suppressed eosinophilia. In addition, it is largely unknown to what extent the few eosinophils remaining after anti-IL5 treatment differ from pre-treatment eosinophils.

The present study is a prospective observational asthma study that aims to use microscopic analysis to investigate the composition and subtypes of blood leukocytes collected before and after instantiated mepolizumab treatment. Comparisons are made to patients already on mepolizumab treatment, asthma patients without any biological treatment, and non-diseased control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma (the asthma patient arms)
* Eligible for Mepolizumab treatment as per the country-specific prescribing information (the arms with Mepolizumab)

Exclusion criteria:

* Any diagnosed infection (all arms)
* Previous history of lung disease, chronic inflammatory condition, atopy, or cardiovascular disease. Diagnosed or perceived infection within 3 weeks prior to blood sampling (Healthy non-asthma control subjects)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All asthma patients will be recruited at the Department of Allergology and Lung Medicine, Skåne University Hospital (SUS), Lund, Sweden. Healthy control subjects are recruited by local advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-18 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Eosinophil Marker Expression | Change from baseline at 1-3 days, 1 week, 4 weeks, and 4 months after initiated biological treatment
  Quantitative immunohistochemical analysis of eosinophil marker expression in blood leukocyte pellets
Change in Blood Basophil Marker Expression | Change from baseline at 1-3 days, 1 week, 4 weeks, and 4 months after initiated biological treatment
  Quantitative immunohistochemical analysis of basophil marker expression in blood leukocyte pellets
Change in Blood Leukocyte Composition | Change from baseline at 1-3 days, 1 week, 4 weeks, and 4 months after initiated biological treatment
  Immunohistochemical determination of the relative proportion (percent) of the leukocyte populations in blood leukocyte pellets

SECONDARY OUTCOMES:
Change in Blood T Lymphocyte Marker Expression | Change from baseline at 1-3 days, 1 week, 4 weeks, and 4 months after initiated biological treatment
  Quantitative immunohistochemical analysis of T lymphocyte marker expression in paraffin-embedded blood leukocyte pellets
Change in Blood B Lymphocyte Marker Expression | Change from baseline at 1-3 days, 1 week, 4 weeks, and 4 months after initiated biological treatment
  Quantitative immunohistochemical analysis of T lymphocyte marker expression in paraffin-embedded blood leukocyte pellets
Leukocyte Total Cell Counts | Change from baseline at 1-3 days, 1 week, 4 weeks, and 4 months after initiated biological treatment
  Routine hemacytometer total leukocyte cell counts

OTHER OUTCOMES:
Change in Forced Expiratory Volume in 1 second (FEV1) | Change from baseline at 4 weeks, and 4 months after initiated biological treatment.
  Spirometry: Forced Expiratory Volume, 1s; (FEV1).
Change in Forced Vital Capacity (FVC) | Change from baseline at 4 weeks, and 4 months after initiated biological treatment.
  Spirometry: Forced Vital Capacity (FVC)
Change in Exhaled FeNo | Before and 1-3 days, 1 week, 4 weeks, and 4 months after initiated biological treatment.
  Fractional exhaled NO will be measured at multiple flows

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Erjefält, Principal Investigator — Lund University Hospital
Locations (1):
- The Lung and Allergy Clinic, Skåne University Hospital (SUS), Lund, Skåne County, Sweden